CLINICAL TRIAL: NCT05051618
Title: Exercise Training for Managing Major Depressive Disorder in Multiple Sclerosis
Acronym: METS in MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert W Motl, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1354; W81XWH2110952 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2021-09-02; First posted 2021-09-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Major Depressive Disorder
Keywords: Multiple Sclerosis; MS; Depression; MDD; Exercise; Physical Activity; Intervention; Behavior
MeSH Terms: conditions — Multiple Sclerosis; Depressive Disorder, Major; Depression; Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POWER-MS (Experimental): The POWER-MS condition will deliver the Guidelines for Exercise in MS (GEMS) program with a remotely coached/guided, home-based setting using telerehabilitation. GEMS recommends 30 minutes of moderate intensity aerobic activity, 3x/week AND strength training exercises for major muscle groups, 3x/week.
  Interventions: Behavioral: POWER-MS
- FLEX-MS (Active Comparator): The FLEX-MS condition will primarily focus on flexibility as the applicable exercise modality. As such, the program will emphasize that flexibility is an important component of fitness. The goal would be for each participant to enhance their flexibility by engaging in a titrated exercise prescription where the number of sets and time to hold per set will increase throughout the 16-week program.
  Interventions: Behavioral: FLEX-MS

INTERVENTIONS:
Behavioral: POWER-MS — The POWER-MS intervention includes both aerobic exercise and resistance exercise:
  Aerobic Exercise:
  The goal of the aerobic exercise training is for participants to achieve three moderate-intensity walking sessions of 30+ minutes per session by the end of the 16-week intervention.
  Resistance Exercise:
  Participants will complete resistance exercise training that consists of 1-2 sets (10-15 repetitions) of 5-10 exercises targeting the lower body, upper body, and core muscle groups performed three days per week, with the sets, repetitions and number of exercises increasing based on an individualized difficulty level.
  Arms: POWER-MS
Behavioral: FLEX-MS — The FLEX-MS intervention is specifically a stretching exercise prescription. All exercise movements are consistent throughout the program. At the beginning of the program, the stretching exercise sessions will take five minutes (1 set) three days per week (15 minutes per week). By the end of the 16-week program, the sessions will take about 30 minutes (2 sets) to be performed three days per week (1.5 hours per week).
  Arms: FLEX-MS

SUMMARY:
The purpose of this research is to examine the effects of two different exercise training regimens for managing depression and improving other health indicators among persons with multiple sclerosis (MS). The project will enroll persons with MS and major depressive disorder (MDD) between 18 and 64 years of age. The investigators will enroll a total of 146 participants.

This is a Phase-II trial that compares the efficacy of an exercise training program (POWER-MS) compared with a stretching program (FLEX-MS) for immediate and sustained reductions in the severity of depression among persons with MS who have MDD.

ELIGIBILITY:
Inclusion Criteria

* Physical confirmed diagnosis of Multiple Sclerosis (MS)
* Diagnosis of Major Depressive Disorder (MDD) - see below (MINI)
* English as primary language
* Eligible age (between 18 and 64 years old)
* Relapse and steroid free in past 30 days
* Internet and email access
* Willingness to complete the testing and questionnaires, wear the accelerometer, undergo randomization, and engage in exercise testing

Exclusion Criteria

* Godin Leisure Time Exercise Questionnaire (GLTEQ): Exclude if health contribution score of 14 units or more. This assessment is administered to confirm insufficient baseline physical activity (i.e., not meeting current PA guidelines)
* Patient Determined Disease Steps (PDDS): Exclude if score above '2' (i.e., greater than mild ambulatory disability). This assessment is administered as the proposed intervention focuses on walking as main modality for exercise training. The scale asks the participant to describe their walking situation on a scale of 0 to 8; where lower scores indicate better walking ability.
* Beck Depression Inventory-Fast Screen (BDI-FS): Exclude if a score less than '4'. The scale measures depression and those with a score of '4' or below likely have very mild depression resulting in floor effects and/or spontaneous remission.
* Physical Activity Readiness Questionnaire (PAR-Q): Exclude if more than one yes/affirmative response on this 7-item self-report assessment. This assessment is administered to exclude those individuals who are at a moderate to high risk for contraindications of injury or possible death when undertaking strenuous or maximal exercise. This is a 7-item self-report tool where more than one yes/affirmative response indicates that an individual is not recommended to engage in physical activity within the capacity of this study. Those scoring more than one yes/affirmative response will be further advised to seek medical guidance before becoming more physically active.
* Telephone Interview for Cognitive Status (TICS-M): Exclude if scores less than 18. This assessment is administered to ensure that all participants can adequately follow directions. The application of the TICS-M is to ensure that participants do not have severe cognitive impairment that might preclude the ability to adhere to the conditions, understand intervention content, and interact with behavior coaches.
* MINI International Neuropsychiatric Interview (version 7.0.2) based on the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V): Include those who meet the criteria for MDD, but exclude for other severe mental illness (obsessive-compulsive disorder, schizophrenia, bipolar or other psychotic disorders) as indicated by the MINI; these persons would require more intensive mental health treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depression Severity (self-report) | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Patient Health Questionnaire (PHQ-9); scores range between 0 (min) and 27 (max), higher scores indicate greater depression severity.
Change in Depression Severity (observer-rated) | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Hamilton Depression Rating Scale (HDRS-17); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of depressive symptoms.

SECONDARY OUTCOMES:
Change in Perception of Fatigue Severity | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Change in Cognitive Performance | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS). The BICAMS includes Symbol Digit Modalities Test (SDMT), first five learning trials of the California Verbal Learning Test-II (CVLT-II), and first three learning trials of the Brief Visuospatial Memory Test-Revised (BVMT-R).
  SDMT scores range between 0 (min) and 110 (max), higher scores indicate better performance.
  CVLT-II scores range between 0 (min) and 80 (max), higher scores indicate better performance.
  BVMT-R scores range between 0 (min) and 36 (max), higher scores indicate better performance.
Change in Quality of Life | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Multiple Sclerosis Impact Scale (MSIS-29); scores range between 0 (min) and 100 (max), higher scores indicate worse quality of life.

OTHER OUTCOMES:
Change in Self-Reported Exercise Behavior | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Godin Leisure Time Questionnaire (GLTEQ); scores range between 0 (min) and 119 (max), higher scores reflect greater levels of physical activity.
Change in Physical Activity | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Accelerometer measured moderate to vigorous physical activity (MVPA) over a seven-day period; scores range between 0 (min) and 1440 (max), higher scores indicate greater physical activity.
Change in Aerobic Capacity | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Aerobic fitness measured as peak oxygen consumption using an incremental exercise test; scores range from 3.5 (min) with no upward bound, higher scores indicate better aerobic fitness.
Change in Muscle Strength | baseline (week 0), immediate follow-up (week 16 or 4 months), and long-term follow-up (week 32 or 8 months)
  Bilateral isometric knee extensor (KE) and flexor (KF) peak torque will be measured using an isokinetic dynamometer; scores range from 0 (min) with no upward bound, higher scores indicate better muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Motl RW, Bombardier CH, Duffecy J, Hibner B, Wathen A, Carrithers M, Cutter G. Study protocol: exercise training for treating major depressive disorder in multiple sclerosis. BMC Neurol. 2024 Apr 17;24(1):131. doi: 10.1186/s12883-024-03634-y. PMID 38632556